CLINICAL TRIAL: NCT00804076
Title: Gene Transfer for Intractable Pain: A Phase I Clinical Trial to Determine the Maximum Tolerable Dose of a Replication-Defective Herpes Simplex Virus Type I (HSV-1) Vector Expressing Human Preproenkephalin (NP2) in Patients With Malignancies
Brief Title: Gene Transfer for Cancer Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diamyd Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP2/P1/07/1
Record Dates: First submitted 2008-12-03; First posted 2008-12-08 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Cancer Pain
Keywords: gene therapy; replication defective HSV vector; pain; enkephalin; intradermal
MeSH Terms: conditions — Cancer Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NP2 (Experimental): Intradermal injection
  Interventions: Biological: NP2

INTERVENTIONS:
Biological: NP2 — Intradermal injection of NP2 at doses ranging from 10e7 to 10e9 pfu at the site of pain.

SUMMARY:
The primary purpose of this study is to examine the safety of NP2 (a nonreplicating HSV-based vector expressing enkephalin) in patients with cancer pain. The secondary purpose is to evaluate efficacy.

DETAILED DESCRIPTION:
Therapeutic HSV-based vectors deliver genes from skin inoculation to sensory neurons to interrupt pain signaling at the spinal level. Side effects may be limited by the focal distribution of vector delivery and preproenkephalin expression. Preproenkephalin is a natural human gene that produces peptides that bind to opioid receptors in the body. The therapeutic being evaluated, NP2, is a replication defective herpes simplex type 1 virus (HSV-1) modified to express the human preproenkephalin gene that has demonstrated efficacy in numerous model of pain, including pain caused by cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intractable pain from malignant disease with a 5 year projected survival of less than 25%.
2. Female patients of childbearing potential who have a negative pregnancy test and using birth control.
3. Patients who have not received recent treatment with a radiation, chemotherapeutic or immunotherapeutic agent and are not expected to undergo such treatment 28 days after injection of NP2.
4. Patients who have not had surgical stabilization/resection within 4 weeks of Screening and have no plans for additional surgical procedures.
5. Patients with adequate bone marrow function, IgG levels greater than 565 mg% and CD4 count greater than 500. .

Exclusion Criteria:

1. Patients with serious uncontrolled medical conditions other than malignancy.
2. Patients with severe liver or renal impairment
3. Patients currently or previously with positive serology for HIV, Hepatitis B or Hepatitis C.
4. Patients with a hemoglobin <9 gm% or uncontrolled coagulopathy or bleeding diathesis.
5. Patients with a clinical diagnosis of any active herpes infection within the past 6 months.
6. Patients who have been vaccinated to prevent HSV infection or a history of shingles or the presence of active shingles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety measured by vital signs, physical exam findings, clinical laboratory analyses and treatment related Adverse Events (AE). | 4 Months

SECONDARY OUTCOMES:
Evaluate changes in cancer-related pain | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: David J Fink, MD, Principal Investigator — University of Michigan Department of Neurology
Locations (5):
- United States (5):
  - Advanced Pharma CR, Miami, Florida
  - Louisiana Research Associates, New Orleans, Louisiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Pain Research of Oregon, LLC, Eugene, Oregon

REFERENCES:
- [Background] Goss JR, Mata M, Goins WF, Wu HH, Glorioso JC, Fink DJ. Antinociceptive effect of a genomic herpes simplex virus-based vector expressing human proenkephalin in rat dorsal root ganglion. Gene Ther. 2001 Apr;8(7):551-6. doi: 10.1038/sj.gt.3301430. PMID 11319622
- [Background] Hao S, Mata M, Goins W, Glorioso JC, Fink DJ. Transgene-mediated enkephalin release enhances the effect of morphine and evades tolerance to produce a sustained antiallodynic effect in neuropathic pain. Pain. 2003 Mar;102(1-2):135-42. doi: 10.1016/s0304-3959(02)00346-9. PMID 12620604
- [Background] Goss JR, Harley CF, Mata M, O'Malley ME, Goins WF, Hu X, Glorioso JC, Fink DJ. Herpes vector-mediated expression of proenkephalin reduces bone cancer pain. Ann Neurol. 2002 Nov;52(5):662-5. doi: 10.1002/ana.10343. PMID 12402268
- [Background] Glorioso JC, Fink DJ. Herpes vector-mediated gene transfer in the treatment of chronic pain. Mol Ther. 2009 Jan;17(1):13-8. doi: 10.1038/mt.2008.213. Epub 2008 Oct 7. PMID 18841093